CLINICAL TRIAL: NCT06346054
Title: Molecular Assessment for Gastro-Esophageal Cancer
Acronym: MAGEC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Stijn Vanstraelen, Principal investigator, Universitaire Ziekenhuizen KU Leuven
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: s68669
Record Dates: First submitted 2024-03-23; First posted 2024-04-03 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Esophageal Cancer; Gastric Cancer; Barrett Esophagus
Keywords: Oncometabolites; Early-stage cancer; Diagnostic testing; Screening
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Barrett Esophagus; Neoplasms | interventions — Breath Tests; Hematologic Tests

STUDY DESIGN:
Intervention Model Description: Participants with gastro-esophageal cancer, participants with Barrett's esophagus and Healthy controls will be monitored in parallel to identify oncometabolic biomarkers related to cancer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gastro-esophageal cancer group (Experimental): Participants with gastroesophageal cancer providing a breath and blood sample for biomarker identification
  Interventions: Diagnostic Test: Breath analysis; Diagnostic Test: Blood analysis
- Barrett's esophagus group (Active Comparator): Participants with Barrett's esophagus providing a breath and blood sample for biomarker identification
  Interventions: Diagnostic Test: Breath analysis; Diagnostic Test: Blood analysis
- Healthy controls (Active Comparator): Healthy controls providing a breath and blood sample for biomarker identification
  Interventions: Diagnostic Test: Breath analysis; Diagnostic Test: Blood analysis

INTERVENTIONS:
Diagnostic Test: Breath analysis — Detection of proteins and volatile organic compounds (oncometabolites) in the exhaled breath
Diagnostic Test: Blood analysis — Detection of proteins and circulating tumor DNA (oncometabolites) in the peripheral blood

SUMMARY:
The goal of this minimally invasive interventional study is to learn if oncometabolic biomarkers, detected in the exhaled breath and blood can identify early-stage gastro-oesophageal cancer in patient at risk for gastro-oesophageal cancer.

The main questions this study aims to answer:

Are oncometabolites proficient and reproducible enough to function as diagnostic biomarkers? Can these biomarkers identify early-stage gastro-esophageal cancer? Researchers will compare participants with gastro-oesophageal cancer to healthy controls and participants with Barrett's esophagus to detect meaningful differences between the groups.

Participants will provide a breath and blood sample during their routine standard of care visits.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any breath or blood analysis
2. >18 years old
3. Barrett's esophagus or treatment naïve gastro-esophageal cancer stage I to IV
4. Voluntary healthy controls

Exclusion Criteria:

1. <18 years old
2. Patient has history of:

   1. Active other cancer than gastro-esophageal cancer
   2. Prior cancer treated <3 years ago
   3. Hepatic dysfunction/liver failure (MELT >7)
3. Any disorder, which in the investigator's opinion might jeopardise participant's safety or compliance with the study plan.
4. Insufficient/unreliable quality of breath (e.g., breath flow) or plasma sample (e.g., haemolytic sample)
5. Incarcerated individuals

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Identification of the concentrations of oncometabolites | year 1-2
  Identify the concentrations of cancer-related metabolites (oncometabolites) in the exhaled breath and blood compared to healthy controls

SECONDARY OUTCOMES:
Assessment of incidence of early-stage cancer | year 2-5
  Distinguish early-stage gastro-oesophageal cancer from Barrett's esophagus and healthy controls based on sensitivity, specificity and accuracy of the oncometabolite concentration
Assessment of incidence of therapy response | year 2-5
  Predict and assess therapy response prior to surgery, based on sensitivity, specificity and accuracy of the oncometabolite concentration
Assessment of percentage change of therapy response | year 2-5
  Assess changes in the concentrations of the oncometabolites related to treatment.
Assessment of incidence of recurrence | year 2-5
  Predict and assess recurrence, based on sensitivity, specificity and accuracy of the oncometabolite concentration

CONTACTS AND LOCATIONS:
Overall Officials: Stijn Vanstraelen, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Philippe Nafteux, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request with the principal investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code